CLINICAL TRIAL: NCT05526391
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous TAK-341 in Subjects With Multiple System Atrophy
Brief Title: A Study of TAK-341 in Treatment of Multiple System Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAK-341-2001; 2022-000336-28 (EudraCT Number); jRCT2011220029 (Registry Identifier: jRCT); 2023-509876-40-00 (EU CTIS Number)
Record Dates: First submitted 2022-09-01; First posted 2022-09-02 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Multiple System Atrophy
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Early PK Cohort: TAK-341 (Experimental): Participants will be randomized to receive TAK-341 at 4-week intervals for up to 52 weeks.
  Interventions: Drug: TAK-341
- Early PK Cohort: Placebo (Placebo Comparator): Participants will be randomized to receive placebo at 4-week intervals for up to 52 weeks.
  Interventions: Drug: Placebo
- Main Cohort: TAK-341 (Experimental): Participants will be randomized to receive TAK-341 at 4-week intervals for up to 52 weeks.
  Interventions: Drug: TAK-341
- Main Cohort: Placebo (Placebo Comparator): Participants will be randomized to receive placebo at 4-week intervals for up to 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-341 — TAK-341 IV infusion
  Other Names: MEDI1341
  Arms: Early PK Cohort: TAK-341; Main Cohort: TAK-341
Drug: Placebo — TAK-341 placebo-matching IV infusion
  Arms: Early PK Cohort: Placebo; Main Cohort: Placebo

SUMMARY:
The main aim is to see how TAK-341 works after 52 weeks in participants with multiple system atrophy as measured by the Unified Multiple System Atrophy Rating Scale Part I (UMSARS).

The study will enroll approximately 138 patients. Participants will receive a total of 13 intravenous infusions every 4 weeks approximately, these may be either of TAK-341 or placebo, after each infusion some blood samplings will be taken and other assessments completed.

This trial will be conducted in North America, Europe and Asia.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-341. The study will evaluate the efficacy, safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of intravenous (IV) TAK-341 in participants with multiple system atrophy (MSA).

The study will enroll approximately 138 participants. The study comprises a screening period of up to 42 days (6 weeks), a 52-week double-blind treatment period, and a follow-up safety visit. Participants will be randomly assigned (by chance, like flipping a coin) to one of the treatment schedules-which will remain undisclosed to the participant, care provider and investigator during the study:

* Early PK Cohort: TAK-341
* Early PK Cohort: Placebo
* Main Cohort: TAK-341
* Main Cohort: Placebo

The change from baseline in UMSARS will be measured at Week 52 post-dose.

This multi-center trial will be conducted worldwide. The duration of treatment in this study will be 52 weeks. Participants will make a follow-up visit to the site after approximately 90 days after the last dose of study treatment.

ELIGIBILITY:
Inclusion criteria:

Diagnostic:

1. The participant has a diagnosis of possible or probable MSA using the modified Gilman et al, 2008 diagnostic criteria.
2. The participant's onset of first MSA symptoms occurred ≤4 years before screening, as assessed by the investigator.
3. Evidence of MSA specific symptoms and deficits as measured by the UMSARS scale.

Exclusion criteria:

Medical History:

1. The participant has any contraindication to study procedures.

Diagnostic Assessments:

1. Presence of confounding diagnosis and/or conditions that could affect participant's safety during the study per investigator judgement.
2. The participant's participation in a previous study of a disease-modifying therapy (with proven receipt of active treatment) will compromise the interpretability of the data from the present study, per consultation with medical monitor or designee.

Other:

1. The participant has participated in another study investigating active or passive immunization against α-synuclein (αSYN) for progressive disease (PD) or MSA, or has had immunoglobulin G therapy, within 6 months before screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in a Modified Unified Multiple System Atrophy Rating Scale (UMSARS) Part I at Week 52 | Up to 52 weeks
  UMSARS Part I (historical review) is a 11-item scale that was adapted from the Unified Parkinson's Disease Rating Scale (UPDRS) and is used to assess activities related to motor disability and related to autonomic dysfunction. Each item is scored from 0 (normal) to 3 (severe). The total score is a sum of scores from all domains and can range from 0 to 33. Higher scores mean poorer health.

SECONDARY OUTCOMES:
Change From Baseline in 11-item UMSARS at Week 52 | Up to 52 weeks
  The 11- item UMSARS includes 11 items from Part I and II to assesses both motor and autonomic disability. UMSARS Part I (historical review) is used to assess activities related to motor disability and autonomic dysfunction. UMSARS Part II (motor examination) is used to measure the functional impairment and specific parkinsonian or cerebellar features. Each item is scored from 0 (normal) to 4 (severe). The total score is a sum of scores from all domains and can range from 0 to 44. Higher scores mean poorer health.
Change From Baseline in UMSARS Total Score (UMSARS Part I + Part II) at Week 52 | Up to 52 weeks
  UMSARS total scale consists of all items from UMSARS Parts I and II. UMSARS Part I (historical review): 12-item scale used to assess activities related to motor disability and autonomic dysfunction. Each item is scored from 0 (normal) to 4 (severe). UMSARS Part II (motor examination): 14-item scale used to measure the functional impairment (eg, speech, rapid alternating movements of the hands, finger taps, leg agility) of selected complex movements, and specific parkinsonian (tremor at rest) or cerebellar (ocular motor dysfunction, heel-shin test) features. Each item is scored from 0 (normal) to 4 (severe).
Change From Baseline in UMSARS Part I at Week 52 | Up to 52 weeks
  UMSARS Part I (historical review) is a modified 11-item scale that was adapted from the UPDRS and is used to assess activities related to motor disability (first 8 items) and 4 novel items related to autonomic dysfunction. Each item is scored from 0 (normal) to 4 (severe). The total score is a sum of scores from all items and can range from 0 to 44. Higher scores mean poorer health.
Change From Baseline in UMSARS Part II at Week 52 | Up to 52 weeks
  UMSARS Part II (motor examination) is a 14-item scale. Most of the items (e.g., speech, rapid alternating movements of the hands, finger taps, leg agility) measure the functional impairment of selected complex movements, and only a few items directly refer to specific parkinsonian (tremor at rest) or cerebellar (ocular motor dysfunction, heel-shin test) features. The motor examination section of UMSARS was based on modified UPDRS-III items in addition to novel items such as heel-knee-shin ataxia. Each item is scored from 0 (normal) to 4 (severe). The total score is a sum of scores from all items and can range from 0 to 56. Higher scores mean poorer health.
Clinical Global Impression-Severity (CGI-S) Score | Up to 52 weeks
  The CGI-S is used to assess the clinician's impression of the participant's clinical condition. The clinician should use his or her total clinical experience with this participant population and rate the current severity of the participant's illness on a 7-point scale ranging from 1 for normal, not at all ill to 7 for among the most extremely ill participants. Higher scores mean better health.
Change From Baseline in Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction (SCOPA-AUT) Total Score | Up to 52 weeks
  The SCOPA-AUT is a patient-reported outcome that assesses autonomic function. Autonomic function is a critical symptom domain for MSA. The scale is self-completed by participants and consists of 25 items assessing the following domains: gastrointestinal (7 items), urinary (6 items), cardiovascular (3 items), thermoregulatory (4 items), pupillomotor (1 item), and sexual (2 items for men and 2 items for women). The score for each item ranges from 0 (never experiencing the symptom) to 3 (often experiencing the symptom). The total composite score including all domains will be reported. The score range is 0 (no symptoms) to 69 (highest burden of symptoms).
Overall Survival (OS) | Up to 52 weeks
  OS is defined as time from the first day of study drug administration to death due to any cause.
Change from Baseline on Levels of Cerebrospinal Fluid (CSF) Free Alpha-synuclein (αSYN) | Up to 52 weeks
Cmax: Maximum Observed Serum Concentration for TAK-341 | Pre-dose on Days 1, 29, 57, 85, 169, 253, 337; at multiple timepoints (up to 24 hours) post-dose on Days 1, 57, 85, 169, 337; anytime once on Days 365, 427 or at early termination (Day 57 applicable to only early PK cohorts)
Tmax: Time of First Occurrence of Cmax in Serum for TAK-341 | Pre-dose on Days 1, 29, 57, 85, 169, 253, 337; at multiple timepoints (up to 24 hours) post-dose on Days 1, 57, 85, 169, 337; anytime once on Days 365, 427 or at early termination (Day 57 applicable to only early PK cohorts)
AUCτ: Area Under the Concentration-time Curve During a Dosing Interval in Serum for TAK-341 | Pre-dose on Days 1, 29, 57, 85, 169, 253, 337; at multiple timepoints (up to 24 hours) post-dose on Days 1, 57, 85, 169, 337; anytime once on Days 365, 427 or at early termination (Day 57 applicable to only early PK cohorts)
CSF Concentration of TAK-341 | Pre-dose on Days 1, 85 (applicable to only early PK cohorts), and 365
  Lumbar puncture for CSF sampling will be performed.
Number of Participants With at Least one Adverse Event (AE) | Up to 52 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a participants administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. Data will be reported for number of participants to be analyzed for safety parameters that will include clinically significant abnormal values for clinical laboratory evaluations, vital signs, ECG parameters, physical examination, neurological examination and Columbia-Suicide Severity Rating Scale (C-SSRS).
Number of Participants With Antidrug Antibody | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (7):
  - Quest Research Institute - Alcanza - HyperCore, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Inland Northwest Research, Spokane, Washington
- Medizinische Universitat Graz, Graz, Styria, Austria
- Denmark (2):
  - Bispebjerg Hospital, København NV, Capital
  - Aarhus Universitetshospital, Aarhus N
- Hopitaux de La Timone, Marseille, Bouches-du-Rhone, France
- Germany (9):
  - Klinikum Groshadern, LMU, München, Bavaria
  - Paracelsus-Elena-Klinik Kassel, Kassel, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum der Ruhr-Universitaet Bochum (UKRUB) - St. Josef-Hospital, Bochum, North Rhine-Westphalia
  - Deutsches Zentrum fur Neurodegenerative Erkrankung, Bonn, North Rhine-Westphalia
  - Universitatsklinikum Munster, Münster, North Rhine-Westphalia
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Charite - Universitatsmedizin Berlin, Berlin
- Italy (6):
  - IRCCS San Raffaele Roma, Rome, Lazio
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Azienda Ospedale Universita Padova, Padua, Veneto
  - Azienda Ospedaliera Universitaria OO.RR. San Giovanni di Dio Ruggi dAragona, Salerno
- Japan (6):
  - Chiba University Hospital, Chuo-ku, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kyoto University Hospital, Kyoto, Kyoto
  - The University of Tokyo Hospital, Bunkyo-Ku, Tokyo
  - Medical Hospital of Tokyo Medical and Dental University, Bunkyo-Ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira-Shi, Tokyo
- Portugal (2):
  - Campus Neurologico Senior, Loures, Lisbon District
  - Hospital Pedro Hispano, Senhora da Hora, Porto District
- Spain (6):
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Southampton General Hospital, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/e0316361bd7044cd?idFilter=%5B%22TAK-341-2001%22%5D